CLINICAL TRIAL: NCT02780778
Title: Apatinib Plus Docetaxel as 2nd Line Treatment in Patients With Advanced Non-squamous and Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AHEAD-HBL0001
Record Dates: First submitted 2016-05-03; First posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): Apatinib：500 mg，po，qd； Docetaxel：60mg/m²，vein input 1hour，every 3w
  Interventions: Drug: Apatinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Apatinib — Targeted therapy Apatinib：500 mg，po，qd
  Other Names: YN968D1
Drug: Docetaxel — chemotherapy Docetaxel：60mg/m²，vein input 1hour，every 3w
  Other Names: Taxotere

SUMMARY:
The purpose of this Phase II, Open-label, single arm, exploratory study is to evaluate the efficacy and the safety of Apatinib（500mg/d）with docetaxel (60 mg/m²) in advanced Non-squamous Non-small cell lung cancer after failure of first line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 75 years of age
* Histologically or cytologic confirmed advanced non-squamous and non-small cell lung cancer.
* EGFR mutation testing negative of sensitive mutations
* At least one measurable lesion which has not received radiotherapy (larger than 10 mm in diameter by spiral CT scan)
* Have failed for 1 lines of chemotherapy
* ECOG performance scale 0 - 1.
* Life expectancy of more than 3 months.
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin
* More than 4 weeks after operation or radiotherapy
* More than 4 weeks for cytotoxic agents
* Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥ 90g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, total bilirubin within 1.25×the upper limit of normal(ULN), and serum transaminase≤2.5×the ULN (If liver metastases, serum transaminase≤5×the ULN), serum creatine ≤ 1.5 x ULN, creatinine clearance rate ≥ 50ml/min,
* Signed and dated informed consent.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Received more than one kind of chemotherapy regimens
* NSCLC received other VEGFR inhibitors (except beacizumab) or docetaxel chemotherapy
* Existing therapy related toxicity of prior chemotherapy and/or radiation therapy
* Intercurrence with one of the following: hypertension, coronary artery disease, arrhythmia and heart failure
* Any factors that influence the usage of oral administration
* The center of the tumor invaded local large blood vessels
* Within 4 weeks before the first use of drugs, occurs pulmonary hemorrhage (≥ CTCAE class 2) or other parts' hemorrhage (≥ CTCAE class 3).
* Within 6 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc.
* Less than 4 weeks from the last clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 1 Day

SECONDARY OUTCOMES:
objective remission rate | 1 Day
disease control rate | 1 Day
Quality of life score | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Zhanyu Pan, Master, Principal Investigator — National Clinical Research Center for Cancer of China
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China